CLINICAL TRIAL: NCT01632722
Title: A Randomized Phase II Study of Perioperative Chemotherapy Plus Bevacizumab Versus Postoperative Chemotherapy Plus Bevacizumab in Patients With Upfront Resectable Hepatic Colorectal Metastases (APPROACH)
Brief Title: Perioperative vs Postoperative Chemotherapy + Bevacizumab in Colorectal Cancer, Liver Mets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Joong Bae Ahn, professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0166
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer; Liver Metastasis
Keywords: colorectal cancer, liver metastasis, bevacizumab, perioperative/postoperative chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ArmA (Active Comparator)
  Interventions: Drug: Bevacizumab, mFOLFOX, FOLFIRI
- ArmB (Active Comparator)
  Interventions: Drug: Bevacizumab, mFOLFOX, FOLFIRI

INTERVENTIONS:
Drug: Bevacizumab, mFOLFOX, FOLFIRI — ArmA (postoperative arm)
  Postoperative mFOLFOX or FOLFIRI regimen, every 2weeks for 12cycles Bevacizumab 5mg/kg IV, every 2weeks for 11cycles beginning with cycle 2
  Arms: ArmA
Drug: Bevacizumab, mFOLFOX, FOLFIRI — ArmB (perioperative arm)
  Perioperative CTx mFOLFOX or FOFIRI regimen, every 2 weeks for 6 cycles Bevacizumab 5mg/kg IV, every 2 weeks for 5cycles (cycles 1-5)
  Postoperative CTx mFOLFOX or FOLFIRI regimen, every 2weeks for 6 cycles Bevacizumab 5mg/kg IV, every 2weeks for 5cycles(cycles 8-12)
  Arms: ArmB

SUMMARY:
Early-stage colorectal cancer(CRC)is localized and resectable, but 20% of the patients have metastatic disease at the time of diagnosis and 50% of all patients eventually die of the disease. The most frequent site of colorectal metastases is the liver, which accounts for 30% to 60% of cases. In these patients, the extent of liver disease is the main determinant of survival. Hepatectomy is the only potentially curative therapy for colorectal liver metastases (CLM), but when traditional criteria for resectability were used, only 10% of patients were candidates for surgical resection.

Although adjuvant systemic therapy after resection of primary colorectal tumors is well established, there are relatively few data on the use of postoperative therapy vs. surgery alone in patients who have undergone resection of liver metastases. In this trial, the absolute increase in the 3-year PFS rate with the addition of FOLFOX4 was a modest but significant 9% in patients who had resection (from 33% to 42%; P = .025). For improving survival in patients with CLM, several studies with biologic agents have been tried. The use of bevacizumab, a monoclonal antibody against vascular endothelial growth factor (VEGF), has resulted in increased response rates in patients with stage IV colorectal cancer and improved OS and PFS. In an ongoing phase II trial presented in ASCO 2008, in patients who were potentially curable through resection of liver metastases, perioperative treatment with capecitabine and oxaliplatin (XELOX) plus bevacizumab yielded an overall response rate of 73% with stable disease in 21% and a mean PFS of 27 months. Response to chemotherapy significantly correlated with a prolonged PFS (P < .001).

On the basis of these backgrounds, we designed a phase II study to compare the effectiveness of combination chemotherapy with perioperative or postoperative bevacizumab treatment in patients with CLM.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal adenocarcinoma
* With hepatic metastasis and no evidence of extrahepatic metastasis (the liver metastases must be determined by a hepatic surgeon to be resectable)
* 20~80 years
* ECOG performance status 0 - 1
* Adequate laboratory findings

Exclusion Criteria:

* Prior chemotherapy for metastatic disease
* Prior adjuvant chemotherapy, if administered within 6 months before study entry
* Previous hepatic-directed therapy including hepatic resection and/or ablation, hepatic arterial infusion therapy, or hepatic radiation therapy
* Uncontrolled medical illnesses including medically uncontrolled infection, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months
* Chronic active hepatitis or cirrhosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-06; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
2 years recurrence-free survival (2Y-RFS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea